CLINICAL TRIAL: NCT06307574
Title: Digital Technology to Support Adherence to Hypertension Medications for Older Adults With Mild Cognitive Impairment
Brief Title: bpMedManage: Digital Technology to Support Adherence to Hypertension Medications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Kathleen Insel, Principal Investigator, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00002804
Record Dates: First submitted 2024-02-12; First posted 2024-03-13 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Aging; Mild Cognitive Impairment; Hypertension
Keywords: Digital Health Intervention; Medication Adherence; Mobile Application; Mild Cognitive Impairment; Aging; Hypertension
MeSH Terms: conditions — Cognitive Dysfunction; Hypertension; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Participants will be screened and randomly assigned to either the bpMedManage-S or bpMedManage-P group
Who Masked: Outcomes Assessor
Masking Description: All primary and secondary outcome assessments following the intervention, Week 4, are blinded. One of the supplementary outcome measures following the intervention at Week 12, requires the assessor to know the group assignment. This outcome pertains to their experience in the intervention. The follow-up outcome assessments at Week 12 will be administered by an unblinded assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bpMedManage-S (Experimental): Intervention group will use a smartphone application with medication reminders plus receive education with standardized information on hypertension and antihypertensive medications on the education portal. They will complete immediate outcomes assessment 4 weeks after the beginning of the intervention and follow-up outcomes 12 weeks after the beginning of intervention.
  Interventions: Behavioral: bpMedManage
- bpMedManage-P (Active Comparator): Participants in the bpMedManage-P group will use a smartphone to receive education with standardized information on hypertension and antihypertensive medications on the education portal. They will complete immediate outcomes assessment 4 weeks after the beginning of the intervention and follow-up outcomes 12 weeks after the beginning of intervention.
  Interventions: Behavioral: bpMedManage

INTERVENTIONS:
Behavioral: bpMedManage — In this 16-week RCT, a total of 100 older adults with MCI will be recruited. There are two treatment arms, bpMedManage-S and bpMedManage-P with 50 participants in each arm. Participants randomized into the bpMEDManage-S intervention arm will use a smartphone application with medication reminders plus receive education with standardized information on hypertension and antihypertensive medications on the education portal. Participants in the bpMedManage-P group will use a smartphone to receive education with standardized information on hypertension and antihypertensive medications on the education portal. Both groups will complete baseline assessments followed by 4 weeks of medication adherence monitoring. At the end of the adherence monitoring period, participants will be randomized into one of the two treatment arms. Immediate outcomes will be assessed 4 weeks after beginning of the intervention. Follow-up outcomes will be assessed 12 weeks after the beginning of the intervention.

SUMMARY:
The purpose of the bpMedManage study is to rigorously test the efficacy of a smartphone technology to help improve high blood pressure medication adherence among older adults with mild cognitive impairment (MCI) in a 16-week randomized controlled trial. A total of 100 older adults will be recruited. There will be two treatment arms, bpMedManage-S and bpMedManage-P with 50 participants in each arm. Participants randomized into the bpMEDManage-S intervention arm will use a smartphone application with medication reminders plus receive education with standardized information on hypertension and antihypertensive medications on the education portal. Participants in the bpMedManage-P group will use a smartphone to receive education with standardized information on hypertension and antihypertensive medications on an education portal. Both groups will complete baseline assessments followed by 4 weeks of medication adherence monitoring. At the end of the adherence monitoring period, participants will be randomized into one of the two treatment arms. Immediate outcomes on primary and secondary measures will be assessed 4 weeks after beginning of the intervention. Follow-up outcomes will be assessed 12 weeks after the beginning of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60+
2. Community-dwelling older adults
3. Self-reported fluent in English
4. Adequate self-reported visual and hearing ability
5. Self-reported memory, thinking, or concentration challenges
6. Self-manage at least one prescribed antihypertensive medication
7. Have and use a smartphone
8. No self-reported history of major depression or other mental health diagnoses
9. No self-reported diagnosis of dementia or other neurological disorder such as stroke, TBI, and Parkinson's disease
10. TICS-M score between 27-37 and Montreal Cognitive Assessment (MoCA) score between 20-26
11. Willing to participate in the study for at least 4 months

Exclusion Criteria:

1. Diagnosis of dementia
2. Lives in assisted living facility or skilled nursing facility

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in medication adherence measured by the Medication Event Monitoring System (MEMS® Cap) | Week 4, Week 12
  A device used to monitor medication adherence. The medication event monitoring system (MEMS) is a cap that fits on medication bottles and records the time and date each time the bottle is opened. Adherence data by MEMS® monitoring will be downloaded to a study laptop from all participants' MEMS® Cap via a USB connected MEMS® cap reader/communicator.
Change in self-reported medication adherence measured by the Medication Adherence Report Scale-5 (MARS-5© Professor Rob Horne) | Week 4, Week 12
  5 items on a 5-point rating scale to assess participant's medication adherence, with lower scores indicating a lower level of adherence.

SECONDARY OUTCOMES:
Change in Systolic and/or Diastolic blood pressure, as measured by taking blood pressure readings | Week 4, Week 12
  Force of blood pushing against blood vessels while the heart beats.
Change in hypertension knowledge measured by the Hypertension Knowledge-Level Scale | Week 4, Week 12
  22-items scale (range: 0-22) with items associated with hypertension, 6 sub-dimensions, and a lower composite score indicating lower knowledge on hypertension.
System Usability measured by the System Usability Scale | Week 4, Week 12
  Scale (range: 0-100) measures one's perceived usability of a system, with lower scores indicating poor system usability.

OTHER OUTCOMES:
Opinion Interview | Week 12
  Understand participant opinions' regarding facilitators and barriers to using the system.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Insel, PhD, Principal Investigator — University of Arizona; Raksha Mudar, PhD, Principal Investigator — University of Illinois, Urbana-Champaign
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - University of Illinois, Urbana-Champaign, Champaign, Illinois

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Aardex Group. (n.d.). MEMS® Button Medication Event Monitoring System. https://aardexgroup.com/about-us/
- [Background] Al-Saleh S, Lee J, Rogers W, Insel K. Translation of a Successful Behavioral Intervention to a Digital Therapeutic Self-Management System for Older Adults. Ergon Des. 2024 Apr;32(2):5-13. doi: 10.1177/10648046211066409. Epub 2022 Feb 24. PMID 38487251
- [Background] Erkoc SB, Isikli B, Metintas S, Kalyoncu C. Hypertension Knowledge-Level Scale (HK-LS): a study on development, validity and reliability. Int J Environ Res Public Health. 2012 Mar;9(3):1018-29. doi: 10.3390/ijerph9031018. Epub 2012 Mar 22. PMID 22690180
- [Background] Brooke, J. (1996). SUS: A quick and dirty usability scale. Usability Evaluation in Industry, 189, 4-7.
- [Background] Chan AHY, Horne R, Hankins M, Chisari C. The Medication Adherence Report Scale: A measurement tool for eliciting patients' reports of nonadherence. Br J Clin Pharmacol. 2020 Jul;86(7):1281-1288. doi: 10.1111/bcp.14193. Epub 2020 May 18. PMID 31823381
- [Background] Insel KC, Einstein GO, Morrow DG, Koerner KM, Hepworth JT. Multifaceted Prospective Memory Intervention to Improve Medication Adherence. J Am Geriatr Soc. 2016 Mar;64(3):561-8. doi: 10.1111/jgs.14032. PMID 27000329
- [Background] Masterson Creber RM, Maurer MS, Reading M, Hiraldo G, Hickey KT, Iribarren S. Review and Analysis of Existing Mobile Phone Apps to Support Heart Failure Symptom Monitoring and Self-Care Management Using the Mobile Application Rating Scale (MARS). JMIR Mhealth Uhealth. 2016 Jun 14;4(2):e74. doi: 10.2196/mhealth.5882. PMID 27302310

DOCUMENTS (2):
  • Study Protocol (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT06307574/Prot_000.pdf
  • Informed Consent Form (2023-11-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT06307574/ICF_001.pdf